CLINICAL TRIAL: NCT02917408
Title: Retrospective Study About Primary Biliary Cholangitis During January 2001 to July 2016 at West China Hospital
Status: Completed | Type: Observational
Sponsor: Xiaoli Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoli Fan, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: PBC-1
Record Dates: First submitted 2016-09-06; First posted 2016-09-28 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Cholangitis; Liver Cirrhosis, Biliary; Cholestasis; Liver Diseases; Liver Cirrhosis; Bile Duct Diseases
MeSH Terms: conditions — Cholangitis; Liver Cirrhosis, Biliary; Cholestasis; Liver Diseases; Liver Cirrhosis; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary biliary cholangitis during January 2001 to July 2016

SUMMARY:
Retrospective study of all patients diagnosed with primary biliary cholangitis during January 2001 to July 2016 at West China Hospital by review of medical records. The following variables will be retrospectively studied: age, sex, first symptoms, clinical characteristics, pathology, treatment, stage, complications of cirrhosis, other autoimmune diseases and long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of PBC at West China Hospital during January 2001 to July 2016.

Exclusion Criteria:

* Simultaneously diagnosed of autoimmune hepatitis or primary sclerosing cholangitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with primary biliary cholangitis during January 2001 to July 2016 at West China Hospital by review of medical records.
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Description of demographics, management patterns (clinical and diagnostic), comorbidities of PBC patients at diagnosis during the past 16 years. | Up to 16 years.

SECONDARY OUTCOMES:
Evaluation of adverse outcome free survival of the PBC cohort during the 16 years. | Up to 16 years.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital,Chengdu, Sichuan, China
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided